CLINICAL TRIAL: NCT00490360
Title: Neoadjuvant Chemotherapy for Resectable Cancer of the Pancreatic Head
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-2001
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Cancer of the Pancreatic Head
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gemcitabine / Cisplatin

SUMMARY:
Neodajuvant chemotherapy with gemcitabine / cisplatin is applied to patients with resectable cancer of pancreatic head.

DETAILED DESCRIPTION:
Neodajuvant chemotherapy with gemcitabine / cisplatin is applied to patients with resectable cancer of pancreatic head. Two cycles of chemotherapy are given on day 1 and 15 each. After restaging excludes disease progression, a standard Whipple procedure is performed.

Staging and restaging procedures include abdominal CT, diagnostic laparoscopy, PET/CT, tumor markers (CEA, CA 19-9) and assessment of the quality of life by the QLQ-30.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: - Age > 18 years

* Histologically or cytologically confirmed resectable ductal adenocarcinoma of the pancreatic head
* WHO-performance status 0-2
* Written informed consent
* Discussion in an intrdisciplinary conference

Exclusion criteria: - Insufficient renal function (calculated creatinin clearance < 60ml(min)

* Insufficient hematologic function (neutrophil count <1'000/ul, platelets < 100'000/ul)
* Uncorrectable coagulopathy
* Severe cholestasis (bilirubin >100mmol/l)
* Distant metastases in liver, lungs or other organs
* Peritoneal carcinomatosis
* Unresectable tumor (s. 4.2.)
* Contraindication for Whipple procedure
* Uncontrolled infection
* Neurotphil count > Â°2
* Estimated life experience < 6 months
* HIV Infection
* Severe medical or psychatric comorbidities which interefere with the participation in this trial or the informed consent
* Female patients in child-bearing age without adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2007 (Actual)
Dates: Start 2001-10; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Resectability rate > 70% after restaging | 2007

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, Department of Surgery, Zurich, Switzerland

REFERENCES:
- [Derived] Heinrich S, Schafer M, Weber A, Hany TF, Bhure U, Pestalozzi BC, Clavien PA. Neoadjuvant chemotherapy generates a significant tumor response in resectable pancreatic cancer without increasing morbidity: results of a prospective phase II trial. Ann Surg. 2008 Dec;248(6):1014-22. doi: 10.1097/SLA.0b013e318190a6da. PMID 19092346